CLINICAL TRIAL: NCT07132034
Title: Study Protocol: Stress Reduction in Breast Cancer Patients During Transition Into Survivorship Using Acupuncture - a Randomized Wait-list-controlled Intervention Study
Brief Title: Stress Reduction Through Acupuncture
Acronym: STREAK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01072;bb21HeinzelmannSch3
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Acupuncture; Breast Cancer; Survivorship
Keywords: Integrative Oncology; Acupuncture; Breast Cancer; Survivorship; Distress
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, non-blinded, two-arm clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture: (Experimental): 8 sessions of acupuncture treatment, once a week
  Interventions: Procedure: Acupuncture
- Wait-listed control group (Placebo Comparator): Supportive care according to local standards will be given which may also include face-to-face psychosocial support or the participation of support groups. 8 weeks after the assessment T1 and upon completion of assessment T2, participants will receive access to 8 sessions of weekly acupuncture treatment.
  Interventions: Other: Standard supportive care

INTERVENTIONS:
Procedure: Acupuncture — 8 sessions of acupuncture treatment (body and auricular acupuncture) will be given once a week after randomization.
  Arms: Acupuncture:
Other: Standard supportive care — Supportive care according to local standards will be given which may also include face-to-face psychosocial support or the participation of support groups
  Arms: Wait-listed control group

SUMMARY:
This randomized controlled trial evaluates whether eight weeks of weekly acupuncture can reduce psychological distress in breast cancer patients who have recently completed primary therapy compared to standard-of-care wait-list control.

DETAILED DESCRIPTION:
Background Psychological distress is common in cancer patients-affecting roughly one-third with diagnosable mental health disorders and about half with significant psychosocial distress. This distress often spikes during diagnosis and treatment, decreases during therapy, but rises again after treatment ends. The transition from active treatment to aftercare is a particularly vulnerable phase, marked by loss of routine medical contact, fear of recurrence, ongoing side effects, and feelings of isolation. In breast cancer survivors, 20-40% experience clinically relevant distress, with many reporting unmet needs for psychological support. Chronic stress in cancer patients is linked to lower quality of life, worse treatment adherence, higher symptom burden, and poorer prognosis.

Acupuncture, a method from traditional Chinese medicine, has shown potential to reduce stress through modulation of the autonomic nervous system-reducing sympathetic overactivation and enhancing parasympathetic activity. It has been shown to improve symptoms such as pain, fatigue, and hot flushes in cancer patients, and to lower stress in other populations. However, there is almost no research on acupuncture's effect on post-treatment stress in breast cancer patients, especially in the critical early aftercare phase. Whether acupuncture can also improve resilience and treatment adherence in this context remains unknown.

Aim of the Study The study aims to investigate whether acupuncture reduces psychological distress in breast cancer patients who have recently completed primary therapy. Specifically, it tests whether the patients receiving acupuncture will have significantly lower perceived stress after eight weeks compared to a wait-list control group. Secondary objectives include exploring the effects of acupuncture on quality of life, fatigue, cognitive function, anxiety, depression, resilience, and therapy adherence, as well as documenting any adverse events.

ELIGIBILITY:
Inclusion criteria:

* Patients with localized breast cancer having completed primary therapy (operation +/- chemotherapy +/- radiotherapy) in the last 6 months - Distress Thermometer ≥ 5 - Age ≥ 18 years - Signed informed consent for participation of the trial
* Prior cancer is allowed
* Prior treatment - including chemotherapy - for a prior malignant tumor (including breast cancer) is allowed
* Concomitant participation in an experimental therapeutic drug trial is allowed
* Ongoing or planned Anti-her2/neu, immune checkpoint inhibitor, antihormonal and CDK4/6 inhibitor therapy or other adjuvant treatment scheduled for > 3 months during study period is allowed
* Use of other complementary methods (including mistletoe) is allowed.

Exclusion criteria:

* Patients with language or cognitive deficits (including impaired consciousness) that are incompatible with the participation in the study
* Severe physical or psychiatric comorbidity that prevents a patient from participating in the study
* Patients incapable of giving consent
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Distress at 8 weeks of intervention | Post-intervention (after completion of the 8 week acupuncture therapy or SOC)
  Distress is assessed after completion of 8 weeks of weekly acupuncture interventions or standard of care (SOC) by the Perceived Stress Scale (PSS-10). PSS-10 is a 10-item questionnaire widely used to assess stress levels in individuals. It measures the degree to which life has been perceived as unpredictable, uncontrollable und overloading over the last month. The responses are rated on a 5-point rating scale with a total score ranging from 0-40 while a higher total score indicating greater stress.

SECONDARY OUTCOMES:
Distress over the course time | Before and after each acupuncture session during the the 8 week intervention period
  Immediate changes in distress before and after the intervention will be assessed over the course of 8 weeks by the Distress Thermometer, a valid and reliable measure developed by the National Comprehensive Cancer Network for screening psychological distress in cancer patients. The German version was adapted by Mehnert et al. A score of 5 or higher at the visual analogue scale. The score ranges from 0-10 while 10 indicates a higher stress level.
Quality of life assessment | Post-intervention (after completion of the 8 week acupuncture therapy or SOC)
  Quality of life is assessed after completion of the 8 week acupuncture therapy or SOC by 30-items EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30). The score ranges from 0-100 while 100 indicates a higher quality of life.
Anxiety | Post-intervention (after completion of the 8 week acupuncture therapy or SOC)
  Anxiety will be measured using the validated questionnaire The Hospital Anxiety and Depression Scale (HADS) for somatically ill patients with good psychometric properties and with satisfactory internal consistency. The scale consists of 14 questions, with each question being assigned a value from 0 to 3. The total score can range from 0 to 21. Scores of 8-10 are considered borderline, 11-15 moderate, and 16 or higher severe anxiety.
Depression | Post-intervention (after completion of the 8 week acupuncture therapy or SOC)
  Depression will be measured using the validated questionnaire The Hospital Anxiety and Depression Scale (HADS) for somatically ill patients with good psychometric properties and with satisfactory internal consistency. The scale consists of 14 questions, with each question being assigned a value from 0 to 3. The total score can range from 0 to 21. Scores of 8-10 are considered borderline, 11-15 moderate, and 16 or higher severe depression.
Resilience | Post-intervention (after completion of the 8 week acupuncture therapy or SOC)
  Resilience is assessed by the Connor-Davidson Resilience Scale 10 (CD-RISC-10). It is the shortened version of a 25-items questionnaire which evaluates the patient's ability to bounce back when diagnosed with a disease. The responses are rated on a 5-point rating scale with the total score ranged from 0-40 while a higher total score indicating greater resilience.
Therapy Adherence | Post-intervention (after completion of the 8 week acupuncture therapy or SOC)
  Adherence to maintenance treatment will be assessed using the Medication Adherence Report Scale-V questionnaire (MARS-V) which consists of 5 items answered on a 5-points-scale. The responses range from 5-25 with higher scores indicating better adherence. Adherence to adjuvant anti-Her2 treatment will be extracted from medical records
Adverse Events: | After each acupuncture session during the the 8 week intervention period
  Adverse events of the acupuncture treatment will be recorded by the acupuncturists using standardized registration sheets at each visit
Fatigue | Post-intervention (after completion of the 8 week acupuncture therapy or SOC)
  Cancer-related fatigue will be assessed using the 13-items Functional Assessment of Chronic Illness Therapy - Fatigue subscale (FACIT-Fatigue). The questionnaire uses 13 items, each scored on a 0-4 Likert scale. The total possible score ranges from 0 to 52, where higher scores indicate less fatigue, and lower scores indicate greater fatigue.
Self-reported cognitive impairment | Post-intervention (after completion of the 8 week acupuncture therapy or SOC)
  Self-reported cognitive impairment will be carried out using the Attention Function Index (AFI), a 13-item questionnaire primarily used for breast cancer patients which measures perceived effectiveness of activities requiring attention. The answers are ranged on a numerical rating scale (0-10) with higher scores indicating better functioning. The AFI has shown correlations with measures of ability to concentrate, cognitive failures, confusion and fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Viola Heinzelmann-Schwarz, Prof.MD, Study Chair — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland